CLINICAL TRIAL: NCT06045962
Title: Effect of Three vs Seven Day Ureteral Stent Removal After Ureteroscopy on Stent Related Symptoms
Brief Title: Optimal Stent Duration After Ureteroscopy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Karen L. Stern, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-011586
Record Dates: First submitted 2023-09-07; First posted 2023-09-21 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Ureteral Stent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Uncomplicated Ureteroscopy and Stent Placement for 3-5 days (Active Comparator): After standard of care ureteroscopic procedure stents will be left indwelling for 3-5 days
  Interventions: Device: Ureteral stent
- Uncomplicated Ureteroscopy and Stent Placement for 7-9 days (Experimental): After standard of care ureteroscopic procedure stents will be left indwelling for 7-9 days
  Interventions: Device: Ureteral stent

INTERVENTIONS:
Device: Ureteral stent — Used to open the ureter and help the kidney drain

SUMMARY:
The purpose of this study is to determine how soon ureteral stents can be safely removed following surgery.

DETAILED DESCRIPTION:
The rationale for this study is to determine if there is a difference in symptoms or complications among patients undergoing uncomplicated ureteroscopy for stone removal with shorter indwelling stent duration. Currently there are only a few small studies exploring the optimal duration of stent placement after stent placement and no multicenter randomized control trials. The investigation aim is to determine if earlier ureteral stent removal will reduce urinary symptoms after stent removal and improve quality of life without increasing risk of negative side effects. Using questionnaires for stent related symptoms the researchers will assess stent indwelling time effect on patient reported side effects.

ELIGIBILITY:
Inclusion Criteria

* Participants undergoing unilateral stone treatment. Patients may have stones present bilaterally, but must only be having unilateral intervention.
* The ureteroscopy must be uncomplicated
* Patients undergoing semi-rigid ureteroscopy only, flexible ureteroscopy only, or a combination

Exclusion Criteria

* Pregnancy
* A stent or nephrostomy tube placed prior to surgery
* Complex ureteroscopy - ureteral injury, ureteral perforation, ureteral stricture, impacted stone
* Infection or struvite stones
* Recurrent Urinary Tract Infection (UTI): 2 culture proven UTI in 6 months or 3 culture proven UTIs in one year
* No stone evident on ureteroscopic evaluation of ureter or kidney
* Transplant kidney
* Variant anatomy (horseshoe, pelvic kidney)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Urinary Symptom Scores | Post-operative day 2-3 and 2-3 days after stent removal
  The urinary symptoms will be assessed using the self-reported Canadian Endourology Group Stent Symptom Score. Seven item questionnaire to assess urinary stent symptoms using a 5-point Likert scale; higher score indicated worse outcome.

SECONDARY OUTCOMES:
Change in Pain Scores | Post-operative day 2-3 and 2-3 days after stent removal
  Pain score as indicated in the self-reported Canadian Endourology Group Stent Symptom Score questionnaire with a scale of 0-10 (10 being the worst)
Change in Quality of life | Post-operative day 2-3 and 2-3 days after stent removal
  Change as calculated using the Wisconsin "Living With Kidney Stones" Questionnaire, which is a validated document assessing the quality of life of kidney stone patients. Likert scale 1-5 on 28 items total score range 28-140, with a lower score being associated with a lower quality of life.
Return to work | 30 days
  Number of days participants return to work
Complications | 30 days
  Number of subjects to experience complications assessed by telephone, epic messages, ER visits related to procedure, unanticipated provider visits, and hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Stern, MD, Principal Investigator — Mayo Clinic
Locations (11):
- United States (9):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - University of California San Diego, San Diego, California
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic Minnesota, Rochester, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University, Nashville, Tennessee
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - University of Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials